CLINICAL TRIAL: NCT00590291
Title: Genetic Studies of Coronary Artery Disease and Arteriovenous Malformation (GeneQuest) Molecular Determinants of Coronary Artery Disease
Brief Title: Molecular Determinants of Coronaruy Artery Disease
Acronym: GeneQuest
Status: Terminated | Type: Observational
Why Stopped: Sequencing completed early
Sponsor: John Barnard (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, John Barnard, PI, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: GeneQuest; IRB4333 (Other: Cleveland Clinic IRB); 1R01HL121358 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease; Arteriovenous Malformations; Myocardial Infarction
Keywords: Coronary Artery Disease; Arteriovenous Malformations; Myocardial Infarction; CAD; MI; Heart Attack; AVM; genetic; familial
MeSH Terms: conditions — Coronary Artery Disease; Arteriovenous Malformations; Myocardial Infarction

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For each participant, 10 ml of blood for lymphoblastoid cell line immortalization, 10-20 ml blood for DNA extraction, or two buccal swabs. If gene identified, blood samples from children to identify the children affected with this gene will be obtained. When available, biopsy tissues for extracting DNA, RNA, protein, or for cell biological studies will be obtained. Human genomic DNA will be prepared from peripheral blood lymphocytes, biopsy tissue, or cell lines derived from Epstein Barr virus transformed lymphocytes 15. DNA will be used for a variety of purposes including linkage analysis and mutational screening.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: premature CAD and MI, AVM
- Controls: No CAD, MI, AVM

SUMMARY:
The purpose of this study is to discover genes that may cause Coronary Artery Disease (CAD) or Arteriovenous Malformation (AVM).

DETAILED DESCRIPTION:
The purpose of this study is to discover genes that may cause Coronary Artery Disease (CAD) or Arteriovenous Malformation (AVM). Many human diseases are inherited or passed from parent to child in families. These diseases occur because of damage to a gene(s), the genetic material that is also called DNA. Scientists can now use modern molecular techniques to locate and to find certain genes within the DNA (genetic material) of a person, and to follow their inheritance in a family. To find these disease-causing genes requires studies of many affected with the disease and their family members. The purpose of this study is to locate and to find the genes for coronary artery disease (CAD) which occurs when one or more of the arteries that carry oxygen-rich blood from your heart to the rest of your body develop blockages; or, arteriovenous malformation (AVM) which causes abnormal vascular connections between arteries and veins, particularly near the heart. Findings of the genes causing CAD and AVM will have far-reaching effect on the diagnosis, treatment, and prevention of coronary artery disease and arteriovenous malformation. These studies will lead to possible genetic diagnosis, early detection of persons at risk for developing CAD or AVM (even in the absence of symptoms), development of effective drugs, more rational and specific therapeutic interventions, treatments and ultimately, prevention of coronary heart disease. Approximately 3-5 years are required to find one human disease gene.

ELIGIBILITY:
Inclusion Criteria:

* Males at least 45 years old and premenopausal females at least 50 years old at the time of onset of any of the following:
* PTCA
* MI
* CABG
* Must have a living sibling meeting the same criteria.

Exclusion Criteria:

* Substance Abuse in the absence of angiographic coronary stenosis
* Congenital Heart Disease

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CAD or AVM and their family members and 500 normal control individuals The total number enrolled is 2,980, and approximately 2,000 recruited at the Cleveland Clinic.
  We will comply with the NIH guidelines by including women and members of minority groups and their subpopulations in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1461 (Actual)
Dates: Start 1995-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Disease | 2009
Arteriovenous Malformation | 2009

SECONDARY OUTCOMES:
Myocardial Infarction | 2009

CONTACTS AND LOCATIONS:
Overall Officials: John Barnard, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States